# Understanding Participation Trends: An Examination of Patients in Hepatic Encephalopathy Clinical Trials

An Informed Consent Form For Power Clinical Trial's Hepatic Encephalopathy Observational Clinical Study

Date: December 29, 2023

Unveiling the Introduction to the Informed Consent Form

This summary aims to present an outline of our observational clinical study, emphasizing its processes, potential risks, and advantages for participants. While your consent is mandatory, your involvement remains voluntary, granting you the right to withdraw without repercussions.

Our study endeavors to comprehend why individuals with hepatic encephalopathy opt to join, continue, or disengage from clinical trials. The main procedures involve completing questionnaires and follow-up calls, designed to minimize any potential risks to participants.

Despite participants not experiencing direct medical benefits in this observational study, the collected data will assist in identifying strategies to enhance clinical trial participation rates, ultimately benefiting those affected by hepatic encephalopathy.

The study's discoveries will provide invaluable insights into the factors influencing clinical trial participation rates. Our objective is to refine recruitment strategies and elevate patient engagement in trials, leading to improved treatment options and outcomes for hepatic encephalopathy patients. Nevertheless, engaging in this study is voluntary, and declining will not impact your rights or privileges.

Thoroughly reviewing the consent form and seeking clarification on any concerns before making a decision are pivotal. Engaging in discussions with family, friends, advisors, and healthcare professionals is recommended to ensure an informed choice.

Participation remains entirely voluntary, granting the freedom to withdraw at any time without facing any adverse effects.

Exploring Factors Influencing Hepatic Encephalopathy Clinical Trial Participation

Clinical trials play a critical role in advancing hepatic encephalopathy treatments, but concerns exist regarding the representation of participants. This study aims to investigate the influences behind patient choices regarding involvement, discontinuation, or re-engagement in hepatic encephalopathy clinical trials. Uncovering these factors is essential to enhance the relevance and efficacy of future research endeavors.

Ensuring a comprehensive analysis, our focus lies on recruiting a diverse demographic. We seek to understand how factors such as age, race, income, and education impact participation decisions. This collected information aims to devise improved strategies for engaging underrepresented groups in upcoming clinical trials.

Participation in this study is voluntary, enabling individuals to withdraw without repercussions. The study procedures, involving completing questionnaires and follow-up calls, pose minimal risks. Prospective participants are strongly advised to review the consent form thoroughly and seek clarification for any uncertainties.

In essence, this trial aims to deepen our understanding of the factors influencing participation in hepatic encephalopathy clinical trials. Elevating participation rates could expedite the development of innovative treatments for this challenging condition.

Analyzing Participation Trends Among Hepatic Encephalopathy Patients in Clinical Trials

Our research aims to deeply understand the underlying factors that influence the decisions made by hepatic encephalopathy patients regarding their involvement in clinical trials—be it enrollment, withdrawal, or completion. We intend to identify possible

participants by leveraging electronic medical records from past or ongoing interventional trials.

Upon expressing interest, participants will receive a comprehensive consent form elucidating the study's objectives and their rights. Data collection will encompass biweekly questionnaires covering demographics, medical history, and factors guiding their involvement. Additionally, we plan to conduct comprehensive quarterly phone or video interviews to gain deeper insights.

The statistical analysis of the accumulated data aims to reveal the diverse factors that shape patient participation in clinical trials. Sharing these findings through conferences and scholarly publications aims to benefit various stakeholders involved in clinical trials.

Our objective is to utilize these findings to improve and fortify future clinical studies for hepatic encephalopathy patients, thereby strengthening recruitment approaches and enhancing retention rates.

Participation in this study remains entirely voluntary, ensuring withdrawal without any adverse consequences. Minimal risks involve questionnaire completion and follow-up interviews. Our research team is readily available to address any queries or concerns.

Evaluating Risks in Hepatic Encephalopathy Observational Studies

Hepatic encephalopathy observational studies do not involve experimental treatments, yet participation may entail potential risks. These risks might encompass breaches in privacy, emotional distress due to the study's nature, and possible negative outcomes from trial-related procedures.

Before participating, it's crucial to thoroughly review and understand the informed consent form and discuss any concerns with the research team. The team will provide detailed information on potential risks, study benefits, and safety measures implemented to safeguard participants' well-being.

Exploring the Potential Benefits of Hepatic Encephalopathy Observational Studies

Participating in observational clinical trials focused on hepatic encephalopathy offers patients the chance to contribute to medical advancements and potentially enhance future treatment choices. Despite the absence of experimental treatments, patients can still receive comprehensive care throughout the study.

Before making a decision about trial involvement, patients should thoroughly evaluate the potential benefits and risks, taking into account their individual situation and goals. Seeking guidance from healthcare professionals and the research team is vital in making an informed choice.

#### Contemplating Aspects Affecting Your Trial Involvement

Understanding that your participation in a clinical trial could be discontinued without your explicit consent is crucial. Researchers or sponsors might end the trial due to reasons such as study suspension, withdrawal of financial support, or if it's deemed beneficial for your welfare.

Moreover, your involvement might cease due to declining health, pregnancy, choosing to withdraw following substantial changes or non-adherence to study guidelines. Deliberating on these factors before committing to a clinical trial is of utmost importance.

## Perspective on Hepatic Encephalopathy Clinical Trials

Participation in hepatic encephalopathy clinical trials remains entirely voluntary, allowing participants the freedom to withdraw without facing negative repercussions.

For a comprehensive overview of <u>hepatic encephalopathy research</u> globally, clinicaltrials.gov, overseen by the National Institutes of Health (NIH), functions as an extensive database of trials. The site enables users to refine their search based on location and specific medical conditions.

Additionally, Power's reference page provides an up-to-date compilation of ongoing <u>hepatic encephalopathy clinical trials</u> currently seeking participants.

Exploring Clinical Trial Diversity Through Online Resources

Numerous online platforms cater to individuals seeking a comprehensive understanding of clinical trial diversity. Here are a couple of articles that may pique your interest:

Gross, Annette S., Anya C. Harry, Christine S. Clifton, and Oscar Della Pasqua.

"Clinical trial diversity: An opportunity for improved insight into the determinants of variability in drug response." *British Journal of Clinical Pharmacology* 88, no. 6 (2022): 2700-2717.

Varma, Tanvee, Cary P. Gross, and Jennifer E. Miller. "Clinical Trial Diversity—Will We Know It When We See It?." *JAMA oncology* (2023).

These resources offer valuable insights into the challenges faced in achieving diversity within clinical trials and suggest potential strategies to address these issues.

#### Upholding Privacy in Research Investigations

Ensuring the confidentiality of the information gathered for this research is our utmost priority. Though complete confidentiality cannot be universally guaranteed, extensive measures are implemented to protect it. Please note that legal obligations might require the disclosure of personal information. However, any research publications or presentations will safeguard your anonymity by refraining from disclosing your name or any personally identifying data.

Various entities, including accrediting bodies, government regulatory authorities (such as the FDA and OHRP), safety monitors, study sponsors, and authorized representatives, may access your medical information for research, quality assurance, and data analysis purposes.

In exceptional cases, we might request an "Authorization Form" delineating the utilization and sharing of your information for this study. Prior to sharing your information or research samples with Power researchers, other university institutions, or external commercial entities for future research, explicit consent will be sought. Rest assured, your confidential data will be handled securely and deleted as appropriate.

## Acknowledgment of Informed Consent Terms

Your signature on this consent agreement indicates your acknowledgment and acceptance of the following terms:

- Complete and comprehensive understanding of this informed consent form, with encouragement to seek alternate perspectives before making a decision.
- Satisfactory clarification of all your queries related to the research project and its methodologies, equipping you with the essential information for study participation.
- Consideration of potential benefits, drawbacks, and alternatives associated with participating in the research.
- Assurance that your voluntary involvement in the research study will not curtail your legal rights.
- Timely communication of any significant updates that might influence your decision to continue participating in the research study.
- Receipt of this consent form, providing you with the opportunity to address any lingering questions.

| Participant's Signature | | |
|---|---|---|
| Name of Participant | Signature of Participant | Date |
| Verification by the Researcher | | |
| • | | |
| In my role as the researcher, I have inquiries and strived to offer a comp reaffirmed that the patient's involven | lete comprehension of the stud | ly. Additionally, I have |
| Signature of Researcher Who I | Received Consent | |
| Name of Investigator | Signature of Investigator | Date |